CLINICAL TRIAL: NCT02044640
Title: Identifiable Factors That May Lead to Postoperative Nausea and Vomiting After Simple Laparoscopic Appendectomy
Status: Withdrawn | Type: Observational
Sponsor: Brian Kenney (Other)
Responsible Party: Sponsor-Investigator, Brian Kenney, General Surgeon, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB13-00480
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Appendectomy: Patients undergoing a laporascopic appendectomy
  Interventions: Procedure: Appendectomy

INTERVENTIONS:
Procedure: Appendectomy

SUMMARY:
This is a retrospective chart review meant to identify any factors that are correlated with and may possibly lead to postoperative nausea and vomiting in order to predict need for longer hospital stays and potentially decrease postoperative nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Simple Appendectomy
* Uncomplicated surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing a laparoscopic appendectomy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Postoperative nausea and vomiting | During 1st 24 hours post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States